CLINICAL TRIAL: NCT03051126
Title: Establishment of a Parathyroid Tissue Bank
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LAB08-0034
Record Dates: First submitted 2017-02-02; First posted 2017-02-13 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Parathyroid Disease
Keywords: Parathyroid disease; Parathyroid Tissue Bank; Database; Blood samples
MeSH Terms: conditions — Parathyroid Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Up to 40cc of blood will be collected from all patients during routine blood draws at follow-up appointments through the care cycle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parathyroid Disease Tissue Bank: Participants scheduled for surgical treatment of parathyroid disease and/or patients with MEN1, and/or those presenting with hyperparathyroidism and/or pancreatic lesion, who are scheduled for pancreas tumor intervention.
  Interventions: Other: Tissue Samples

INTERVENTIONS:
Other: Tissue Samples — Fresh residual tissue samples will be obtained during parathyroid and/or pancreas tumor intervention (for pancreas tumor intervention in MEN1 patients with hyperparathyroidism and pancreatic lesions).

SUMMARY:
To develop a tissue bank library for patients with parathyroid disease who have undergone surgery and/or biopsy, and/or who may undergo surgical intervention at M. D. Anderson Cancer Center or outside centers, and/or all patients seen through the Parathyroid Center at participating sites, whether or not the patients undergo treatment for their disease. The tissue bank will contain both normal parathyroid tissue and diseased tissue, and will provide a resource for the ongoing study of parathyroid disease and management.

DETAILED DESCRIPTION:
Fresh residual tissue samples will be obtained during parathyroid and/or pancreas tumor intervention (for pancreas tumor intervention in MEN1 patients with hyperparathyroidism and pancreatic lesions).

In addition, outside paraffin tissue blocks or slides will be requested from patients presenting to MDACC, or to participating family members who have had prior surgery outside of MD Anderson.

Forty cubic centimeters (40 ccs) of whole blood will be obtained from individuals for peripheral blood lymphocyte, plasma, and serum separation and analysis per event. Collections may be made at any or all of the following timepoints: preoperatively, during intervention, and/or at subsequent follow-up visits for up to fifteen years.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible participants will include patients presenting at MD Anderson Cancer who are scheduled for surgical treatment of parathyroid disease and/or patients with MEN1, and/or those presenting with hyperparathyroidism and/or pancreatic lesion, who are scheduled for pancreas tumor intervention, as well as patients having had surgery and who have had residual tissue stored under LAB02-518, LAB03-0320 or prior front door consents, or who have had surgery at other centers and provide signed authorization to obtain the tissue from the outside institution.
2. In addition, eligible participants may include family members of MD Anderson patients who have been diagnosed with parathyroid disease and who have had surgery at other centers, and who provide a signed authorization to obtain the tissue from outside facilities AND/OR who begin care at MD Anderson and will be having intervention at MD Anderson.

Exclusion Criteria:

N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Tissue bank library for patients with parathyroid disease who have undergone surgery and/or biopsy, and/or who may undergo surgical intervention at M. D. Anderson Cancer Center or outside centers, and/or all patients seen through the Parathyroid Center at participating sites, whether or not the patients undergo treatment for their disease.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2009-07-09 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Tissue Collection Obtained During Parathyroid and/or Pancreas Tumor Intervention to Establish a Tissue Bank Library for Ongoing Study of Parathyroid Disease and Management | 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Nancy D. Perrier, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org